CLINICAL TRIAL: NCT06689176
Title: Chlorhexidine Antiseptic Irrigation of the Bowel Segment During Radical Cystectomy and Urinary Diversion After Chlorhexidine Irrigation in Patients Undergoing Radical Cystectomy
Brief Title: Chlorhexidine Antiseptic Irrigation of the Bowel Segment During Radical Cystectomy and Urinary Diversion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Irrimax Corporation (Industry)
Responsible Party: Principal Investigator, John Sfakianos, Associate Professor of Urology, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-23-00340
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Bladder Cancer; Urinary Tract Infection
Keywords: Bladder Cancer; Radical Cystectomy; Ileal Conduit; Neobladder; Chlorhexidine Gluconate; Irrisept
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: This is single center, open-label study where the participants will be identified from the principal investigator and sub-investigator's clinic. All the participants who meet the study criteria and sign the consent form will be assigned to the study intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients undergoing radical cystectomy with urinary diversion (Experimental): Patients undergoing radical cystectomy and ileal conduit or ileal neobladder will receive Irrisept ® Antimicrobial Wound Lavage as intervention
  Interventions: Device: Irrisept® Antimicrobial Wound Lavage

INTERVENTIONS:
Device: Irrisept® Antimicrobial Wound Lavage — Irrisept® Antimicrobial Wound Lavage is a single-use, manual, self-contained irrigation device comprised of a 450mL bottle of 0.05% Chlorhexidine Gluconate (CHG) in 99.95% Sterile Water for Irrigation, United States Pharmacopeia (USP) and an applicator (labeled Irriprobe®). The solution is aseptically filled in a Blow-Fill-Seal (BFS) bottle. The CHG acts as a preservative to inhibit microbial growth in the solution.

SUMMARY:
This is a single arm, interventional pilot study of using chlorhexidine irrigation intra-operatively and post-operatively among patients undergoing radical cystectomy with urinary diversion. The intervention comprises of using irrigation of ileal conduit or ileal neobladder intra-operatively and then for irrigation of either post-surgery with Irrisept ®. The sterilization of urine will be assessed at 10 days after cystectomy. Incidence of symptomatic urinary tract infections within the 30-day post-operative period will be estimated.

DETAILED DESCRIPTION:
Th research team proposes to increase the rate of sterilization of urine from patients with urinary diversion and reduce the incidence of UTI up to 30 ± 7 days post radical cystectomy and urinary diversion using 50 ± 25ml of Irrisept ® irrigation solution lavage of the bowel segment during surgery for a contact time of 2 minutes. For patients who obtain an ileal conduits irrigation using 50 ± 25ml of Irrisept ® will be performed daily for 10 days +/- 3 days and for those patients obtaining ileal neobladders irrigation using 50 ± 25ml of Irrisept ® will continue for 21 days +/- 7 days. The irrigation will continue for the given time described above as this is usually when stents and catheters are removed.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated availability for the duration of the study, and willingness to comply with all study procedures, including willingness to adhere to twice daily irrigation of neobladder or ileal conduit.
* Male or female, ≥ 18 years of age
* Confirmed diagnosis of bladder cancer
* Candidate for radical cystectomy with urinary diversion
* ECOG performance status of 0-2
* Serum creatinine ≤ 1.5 mg/dL

Exclusion Criteria:

* Has undergone or planned to undergo urinary diversion other than ileal conduit or neobladder.
* Pregnancy or lactation.
* Known allergic reactions to components of the Irrisept irrigating system, chlorhexidine.
* Patient must not have any uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants that have negative urine culture | 30 ± 7 days post radical cystectomy with urinary diversion.
  Negative urine culture will be defined as a colony count of less than or equal to 100000 CFU/ml. The urine sample will be collected by catheterization of the conduit with a 16F Foley catheter, which provides the least number of CFU of bacteria compared to collection from the ostomy bag. Patients with ileal neobladder will give a spontaneously voided urine sample when able or will be obtained from catheterized urine for those who cannot void.
Proportion of participants with incident symptomatic UTI | 30 ± 7 days post radical cystectomy with urinary diversion.
  Proportion of participants with incident symptomatic UTI by 30 ± 7 days post radical cystectomy with urinary diversion. Symptomatic UTI will be defined as a positive urine culture in the presence of fever (≥38°C) with or without associated flank/abdominal pain.

SECONDARY OUTCOMES:
Percentage of urine leak from neobladder/ ileal conduit | 30 ± 7 days post radical cystectomy with urinary diversion
Percentage of patients with sepsis | 30 ± 7 days post radical cystectomy with urinary diversion
  Percentage of patients with sepsis (when the body reacts to an infection) will be assessed. In case >/= 10% of participants experience sepsis, the intervention will be considered unacceptable.
Percentage of symptomatic urinary tract infections | 30 ± 7 days post radical cystectomy with urinary diversion
  Symptomatic urinary tract infection is when a person has positive UTI and has fever and other symptoms including pain when passing urine and pain in the lower belly.

CONTACTS AND LOCATIONS:
Overall Officials: John P Sfakianos, MD, Principal Investigator — Associate Professor of Urology
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose. Any purpose. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (TBD).